CLINICAL TRIAL: NCT00429416
Title: A Phase I/II Study of Llme Treated Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Hematological Malignancies
Brief Title: Research Study to Determine if an Experimental Agent, LLME Can Decrease the Incidence and Severity of Graft-Versus-Host-Disease (GVHD) Following Blood (Hematopoietic) Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04U.115; 2003-68 (Other: CCRRC)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Hematologic Malignancies
Keywords: Hematologic Malignancies; GVHD; Graft-Versus-Host-Disease; LLME; CD34+ stem cell infusions; CD34- fraction; Cyclosporine; Mycophenolate Mofetil; HSCT; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease | interventions — fludarabine; fludarabine phosphate; Cytarabine; Cyclophosphamide; Tacrolimus; Mesna; Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LLME to Decrease GVHD Following HSC T (Experimental): To determine if an experimental agent, LLME, can decrease the incidence and severity of Graft-Versus-Host-Disease (GVHD) following hematopoietic stem cell transplantation (HSCT).
  Interventions: Drug: L-leucyl-L-leucine Methyl Ester (LLME); Drug: Fludarabine; Drug: Cytarabine; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mesna; Biological: Granulocyte Macrophage Colony-Stimulating Factor (GM-CSF); Procedure: Hematopoietic stem cell transplantation (HSCT)

INTERVENTIONS:
Drug: L-leucyl-L-leucine Methyl Ester (LLME) — Infusion of L-leucyl-L-leucine methyl ester (LLME) treated donor white blood cells
  Other Names: LLME
Drug: Fludarabine — Fludarabine 30 mg/m2 prior to HSCT infusion
  Other Names: fludarabine phosphate; Fludara
Drug: Cytarabine — Cytarabine 2gm/m2 prior to HSCT infusion
  Other Names: cytosine arabinoside; Ara-C; Arabinofuranosyl Cytidine
Drug: Cyclophosphamide — Cyclophosphamide 1gm/m2 prior to HSCT infusion
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Tacrolimus — Tacrolimus given before and after HSCT infusion
  Other Names: FK-506; Fujimycin
Drug: Mesna — Mesna 1gm/m2/day given prior to HSCT infusion.
  Other Names: Uromitexan; Mesnex
Biological: Granulocyte Macrophage Colony-Stimulating Factor (GM-CSF) — GM-CSF given post HSCT infusion
  Other Names: GM-CSF
Procedure: Hematopoietic stem cell transplantation (HSCT) — CD34 selected allogeneic stem cell infusion with 5x104/kg untreated T cells
  Other Names: HSCT

SUMMARY:
The purpose of this research study is to determine if an experimental agent, LLME can decrease the incidence and severity of Graft-Versus-Host-Disease (GVHD) following blood (hematopoietic) stem cell transplantation

DETAILED DESCRIPTION:
We believe that the risks of allogeneic transplant can be drastically reduced if the following criteria can be met: (1) consistent engraftment, (2) little or no GVHD with the ability to rapidly withdraw immune suppression, (3) rapid recovery of CD4 counts to levels greater than 200 cells/micro liter. Our prior (ongoing) trial attempts to address how LLME treated T cells given as donor lymphocyte infusion (DLI) can address points 2 and 3 above. The current study addresses how treatment of the CD34- fraction of the graft attempts to address points 1 and 2 (and to a lesser extent point 3) above. We believe that if these points can be consistently achieved that the mortality of allogeneic HSCT may be reduced to levels more akin to those of autologous HSCT. We propose to test the hypothesis that LLME-treated T cells will be safe with regard to reducing GVHD or other infusion related toxicities and that their administration as part of the transplant will facilitate engraftment. We believe that this approach will ultimately be an important step in a variety of transplant settings ranging from matched siblings to haplodisparate donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 18 years of age, with no upper age limit.
* Patients must have an ECOG performance status of 0 or 1.
* Any patient with a hematologic malignancy which is unlikely to be cured by conventional treatment is eligible for this study.
* Patients for whom a disease specific protocol exists will be transplanted on those protocols as discussed in the introduction.
* Patients who have had prior autografts may be treated on this protocol.
* Patients must have adequate physical function as measured by the following criteria:
* Cardiac: Asymptomatic or, if symptomatic, then left ventricular ejection fraction at rest must be >40%.
* Hepatic: Aspartate transaminase (AST) micro 3x the upper limits of normal and total serum bilirubin < 2.5 mg/dL. Patients with a higher bilirubin from "benign conditions" such as Gilbert's disease may still be eligible for the study.
* Renal: Serum creatinine within the normal range or if creatinine outside normal range then creatinine clearance > 60 ml/min/1.73m2. Serum creatinine must be less than or equal to 2.0 mg/dl.
* Pulmonary: Asymptomatic or, if symptomatic, DLCO (diffusion capacity) > 45% of predicted (corrected for hemoglobin)
* The patient or guardian(s) must be able to give informed consent to the study.
* Patient must have a suitable donor who is identical for HLA (human leukocyte antigens) -A, -B, -C, -DR. Single antigen mismatches for HLA-A, -B, -C, -DR are also permitted. Donors obtained through the National Marrow Donor Program (NMDP) will follow NMDP guidelines.

Exclusion Criteria:

* Patients who are eligible for a standard myeloablative transplant and for whom a standard myeloablative transplant is preferable will not be treated on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-03; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Wagner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University', Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospital — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- LLME to Decrease GVHD Following HSC T: To determine if an experimental agent, L-leucyl-L-leucine Methyl Ester (LLME), can decrease the incidence and severity of Graft-Versus-Host-Disease (GVHD) following hematopoietic stem cell transplantation (HSCT).
  Treatment Outline:
  Day -6: Fludarabine 30 mg/m2 IV, Cytarabine 2 gm/m2 IV Day -5: Fludarabine 30 mg/m2 IV, Cyclophosphamide 1 gm/m2 IV, Mesna 1 gm/m2 IV Day -4: Fludarabine 30 mg/m2 IV, Cytarabine 2 gm/m2 IV, Mesna 1 gm/m2 IV Day -3: Fludarabine 30 mg/m2 IV, Cyclophosphamide 1 gm/m2 IV, Mesna 1 gm/m2 IV Day -2: Fludarabine 30 mg/m2 IV, Cytarabine 2 gm/m2 IV, Mesna 1 gm/m2 IV Day -1: Rest day Day 0: CD34 selected allogeneic stem cell infusion with 5x104/kg untreated T cells Day 1: Infusion of LLME treated donor CD34 - cells
Period: Overall Study
Arm/Group | LLME to Decrease GVHD Following HSC T
Started | 14
Completed | 13
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | LLME to Decrease GVHD Following HSC T
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.65 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety of CD34+ Stem Cell Infusions Followed by LLME as Measured by 100-Day Mortality
Description: Determine the safety of CD34+ stem cell infusions followed by the LLME treated CD34- fraction. This includes monitoring the patients for any side effects associated with the LLME treated cell infusion or any other unexpected adverse events.
  This regimen will be gauged as to its safety using 100 day mortality as the measured endpoint. Deaths from all causes will be included.
Time Frame: Through 100 days post-transplant or death
Measure: Number; unit: participants
Arm/Group | LLME to Decrease GVHD Following HSC T
Number analyzed (Participants) | 13
participants | 1

2. Secondary Outcome: Rate of Engraftment of Non-Myeloablative Transplants
Description: Determine the engraftment rate of non-myeloablative transplants using CD34+ stem cells and LLME treated CD34- products.
Time Frame: Through 30 days post-transplant
Measure: Number; unit: participants
Arm/Group | LLME to Decrease GVHD Following HSC T
Number analyzed (Participants) | 13
participants | 13

3. Secondary Outcome: Incidence of Grade II-IV Acute Graft-Versus-Host-Disease (GVHD)
Description: Determine the incidence of grade II-IV acute GVHD after administration of grafts when combined with Cyclosporine/Mycophenolate Mofetil for GVHD prophylaxis. GVHD assessments occur daily as an in patient and at each out patient visit.
Time Frame: Through 24 months post-treatment
Measure: Number; unit: participants
Arm/Group | LLME to Decrease GVHD Following HSC T
Number analyzed (Participants) | 13
participants
  Developed grade II-IV GVHD | 3
  Developed cGVHD (Chronic GVHD) | 1

4. Secondary Outcome: Rate of Serious Infectious Complications
Description: Determine the rate of serious infectious complications. A serious infection will be defined as any requiring hospitalization or parenteral therapy.
  CD4 counts will be measured monthly for the first 3 months after transplant.
Time Frame: Through 3 months post-transplant
Measure: Number; unit: participants
Arm/Group | LLME to Decrease GVHD Following HSC T
Number analyzed (Participants) | 13
participants | 2

5. Secondary Outcome: Number of Patients Who Achieve a CD4 Count > 200/Micro-liters
Description: Determine the number of patients who achieve a CD4 count > 200/micro-liters by 60 days after transplant.
Time Frame: Through 60 Days Post Transplant
Measure: Number; unit: participants
Arm/Group | LLME to Decrease GVHD Following HSC T
Number analyzed (Participants) | 13
participants | 13

ADVERSE EVENTS:
Description: "Other Adverse Events" were not collected/assessed
Arm/Group | LLME to Decrease GVHD Following HSC T
Serious Adverse Events (participants affected / at risk) | 10/14
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LLME to Decrease GVHD Following HSC T (N=14)
Diarrhea (General disorders) | 2 (2)
Bone marrow cellularity (General disorders) | 1 (1)
Infection (General disorders) | 3 (7)
Pancyptopenia (General disorders) | 1 (1)
Hematoma (General disorders) | 1 (1)
Death (General disorders) | 7 (7)
Hypersensitivity (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Progressive disease (General disorders) | 1 (1)
Nausea (General disorders) | 3 (3)
Vomiting (General disorders) | 2 (2)
Fevers (General disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Prostatic obstruction (General disorders) | 1 (1)
Pericardial effusion (General disorders) | 1 (1)
Opportunistic infection (General disorders) | 3 (3)
Bladder obstruction (General disorders) | 1 (2)
Hepatic failure (General disorders) | 1 (1)
Renal insufficiency (General disorders) | 1 (1)
Renal failure (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes